CLINICAL TRIAL: NCT03831360
Title: Adaptation and Pilot Study of Yoga to Reduce Depression in Adolescents
Brief Title: Treatments for Improving Mood in Depressed Teens-3
Acronym: TeenThrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1801001977; R34AT009886 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-02-05 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hatha Yoga (Experimental): 12 weeks of hatha yoga
  Interventions: Behavioral: Yoga
- Group CBT (Experimental): 12 weeks of group CBT
  Interventions: Behavioral: Group CBT

INTERVENTIONS:
Behavioral: Yoga — Hatha yoga for depressed adolescents
  Arms: Hatha Yoga
Behavioral: Group CBT — Group cognitive behavioral therapy for depressed adolescents
  Arms: Group CBT

SUMMARY:
Phase 3 is a randomized clinical trial of yoga vs group Cognitive Behavioral Therapy (CBT) for adolescents with depression.

DETAILED DESCRIPTION:
In Phase 3, Study A, the investigators will conduct a pilot Randomized Control Trial (RCT) of 12 weeks of hatha yoga vs. 12 weeks of group CBT.

Participants will be adolescents with depression. Parents will also be invited to participate in assessments regarding their child.

Study B, which will run concurrent to Phase 3, will be for participants who did not meet the depression inclusion criteria or had recent changes in therapy or medications that make them ineligible for Phase 3. Their data will not be analyzed. They are recruited only for group participation.

Participants will be randomized to Phase 3 groups of 12 weeks of hatha yoga or group CBT. Parents will also be invited to participate in assessments regarding their child.

* Due to social distancing requirements related to COVID-19, all interventions have been delivered remotely via video-based platforms as of late March 2020.

ELIGIBILITY:
Inclusion Criteria:

Please note, inclusion criteria for Phase 3 Study A, and Phase 3 Study B are identical, with the exception that, for Phase 3/ Study B, we will not require elevated depressive symptoms (a) or stable treatment (b).

1. Adolescents must have elevated depressive symptoms, defined by a score of 10 or higher on the Quick Inventory of Depression -Adolescent Version-- Clinician Rating (QIDS-A-CR), including endorsement of either sad mood or anhedonia on the QIDS.
2. Other treatment for depression must be stable at baseline. Adolescents do not have to be in other treatment for depression, but, if they are, it must be stable for the past 8 weeks.
3. Adolescents must be aged 13-18.
4. Adolescents must be medically cleared for moderate physical activity by their primary care physician. This criterion may be met by a current (dated in the past year) statement from their pediatrician that the adolescent may participate in school or camp programs including physical education.
5. Adolescents must be able to read and write English sufficient to complete informed consent and engage in interventions.
6. Adolescents aged 13-17 must assent to be in the study, and their parent or legal guardian must consent to their participation. Adolescents aged 18 must consent to be in the study.
7. Able to attend one of the class times.

Exclusion Criteria:

Exclusion criteria for Phase 3 Study A, and Phase 3 Study B are identical.

1. QIDS- A-CR may not be higher than a score of 21. This ensures that adolescents are not severely depressed.
2. Adolescents may not meet criteria for the following:

   * Autism spectrum disorder "cannot be ruled out", and symptoms are of sufficient severity to interfere with study treatment per clinician judgement
   * Current psychotic disorder
   * Lifetime history of a manic episode
   * Anorexia or Bulimia in past 3 months
   * Substance use disorders in past 12 months, and symptoms are of sufficient severity to interfere with study treatment per clinician judgment These will be assessed with the Mini-International Neuropsychiatric Interview (MINI).
3. Adolescents may not have suicide ideation so severe it will interfere with study participation.
4. Adolescents cannot currently be engaged in yoga classes, as this is the study intervention.
5. Adolescents cannot be pregnant as yoga should be modified for pregnancy.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Uebelacker, PhD, Principal Investigator — Butler Hospital; Shirley Yen, PhD, Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available to other researchers upon request.
Supporting Information: Study Protocol, ICF
Time Frame: upon study completion
Access Criteria: PIs will review requests for IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hatha Yoga | Group CBT
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hatha Yoga | Group CBT | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.00 (1.41) | 15.00 (1.46) | 15.00 (1.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 13 | 12 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 11 | 23
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Acceptability is operationalized by the number of participants who attended 8 or more classes out of possible 12. Target was 70% or greater.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 15 | 15
Participants | 11 | 13

2. Primary Outcome: Credibility Expectancy Questionnaire (CEQ) - Credibility Subscale
Description: Credibility assessed with Credibility Expectancy Questionnaire (CEQ), credibility subscale. The credibility subscale of the CEQ, is a 3 item subscale of the 6 item CEQ. The 3 items are each scored on a range of 0-1, and the mean of thise is used in analyses. Higher scores indicate greater credibility.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 14 | 14
score on a scale | 0.72 (.18) | 0.71 (.17)

3. Primary Outcome: Credibility Expectancy Questionnaire (CEQ) - Expectancy Subscale
Description: Patient expectations assessed with the Credibility Expectancy Questionnaire (CEQ), expectancy subscale. The expectancy subscale is a 3 item subscale of the 6 item CEQ. Score ranges from 0-1 and the mean of those scores are analyzed, with higher scores indicating greater expectations.
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 14 | 14
score on a scale | 0.57 (.20) | 0.55 (.24)

4. Primary Outcome: The Client Satisfaction Questionnaire (CSQ-8)
Description: Satisfaction with treatment assessed with The Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item measure with each item measured on a 1-4 scale, and total score range from 8-32. Higher scores indicate greater client satisfaction.
Time Frame: Post intervention (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 9 | 13
score on a scale | 26.8 (4.18) | 26.1 (5.00)

5. Primary Outcome: Home Practice Questionnaire
Description: Number of participants who met criteria for home practice (target of two practices per week) as assessed with a home practice questionnaire.
Time Frame: Post intervention (month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 14 | 15
Participants | 3 | 8

6. Primary Outcome: Systematic Assessment of Treatment-emergent Events-general Inquiry (SAFTEE)
Description: Participant safety/adverse events will be measured using the SAFTEE. Participants will also be asked weekly if they experienced any injuries as a result of yoga.
Time Frame: Post intervention (month 3)
Measure: Count of Participants; unit: Participants
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

7. Secondary Outcome: Quick Inventory of Depression - Adolescent Version - Clinician Rating (QIDS-A-CR)
Description: Change in depression symptom severity will be assessed via blind evaluator using the the QIDS. The QIDS is a 17 item measure with scores ranging from 0-30. Higher scores indicate greater depressive symptoms.
Time Frame: Baseline to post intervention (month 3)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hatha Yoga | Group CBT
Number analyzed (Participants) | 12 | 13
score on a scale | 6.92 (5.20) | 8.23 (3.17)

ADVERSE EVENTS:
Time Frame: Three months
Arm/Group | Hatha Yoga | Group CBT
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hatha Yoga (N=15) | Group CBT (N=15)
flu (Immune system disorders) | 1 (1) | 2 (2) — flu or mild COVID related symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03831360/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03831360/ICF_001.pdf